CLINICAL TRIAL: NCT04527731
Title: Fit for Two - A Pilot Study on Physical Activity Levels During Pregnancy
Brief Title: Physical Activity Level During Pregnancy
Acronym: Fit4Two
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Other Study IDs: BB002/20
Record Dates: First submitted 2020-06-17; First posted 2020-08-26 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Physical Activity; Well-being
Keywords: Pregnancy; Physical activity; Accelerometry
MeSH Terms: conditions — Motor Activity | interventions — Accelerometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Accelerometry — Participants are asked to wear an accelerometer during the day for a period of seven days.

SUMMARY:
This study examines (1) the extent and intensity of physical activity among women in different phases of their pregnancy and (2) the relationship between patterns of physical activity in pregnancy and well-being.

DETAILED DESCRIPTION:
This study examines physical activity in different phases of pregnancy using accelerometry. The recruitment of pregnant women (N=30) in the first or second trimester (until week 23) will be realized over different channels (e.g, local newspapers, facebook, and leaflets in gynecological practices, shopping centers, and nurseries).

Informed consent consists of: (i) activity recording over seven consecutive days using an accelerometer, (ii) completion of standardized questionnaires, (iii) participation in a cardiac ultrasound examination in the German Center for Cardiovascular Research (DZHK) - examination center.

Participants are asked to wear an accelerometer at daytime, and over seven consecutive days, in trimester 1 (week 9-12), trimester 2 (week 23-26), and trimester 3 (week 36-39). Women who are attended the study in the first trimester wear the device up to three time whereas those who are attended the study in their second trimester wear the device up to twice. At the end of each measurement period women are invited to fill in a self-administered questionnaire. Also they are invited to participate in a cardiac ultrasound examination. Optionally, participants may receive feedback on their physical activity measured by accelerometer as well as about results of cardiac ultrasound examination upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

- current pregnancy, until pregnancy week 23

Exclusion Criteria:

* cognitive impairment
* insufficient language skills

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience Sample (female only)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Extent and intensity of physical activity between pregnancy week 9 and 12 | between pregnancy week 9 and 12
  Assessement via accelerometry
Extent and intensity of physical activity between pregnancy week 23 and 26 | between pregnancy week 23 and 26
  Assessement via accelerometry
Extent and intensity of physical activity between pregnancy week 36 and 39 | between pregnancy week 36 and 39
  Assessement via accelerometry

SECONDARY OUTCOMES:
Well-being | between pregnancy week 9 and 12
  Assessement via self-administered questionnaire: The World Health Organisation- Five Well-Being Index (WHO-5),The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Well-being | between pregnancy week 23 and 26
  Assessement via self-administered questionnaire: The World Health Organisation- Five Well-Being Index (WHO-5),The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Well-being | between pregnancy week 36 and 39
  Assessement via self-administered questionnaire: The World Health Organisation- Five Well-Being Index (WHO-5),The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Mother-child bond | between pregnancy week 9 and 12
  Assessement via self-administered questionnaire: Maternal Antenatal Attachment Scale (MAAS) consists of 19 items which are scored 1-5, with higher scores indicating higher levels of bonding.
Mother-child bond | between pregnancy week 23 and 26
  Assessement via self-administered questionnaire: Maternal Antenatal Attachment Scale (MAAS) consists of 19 items which are scored 1-5, with higher scores indicating higher levels of bonding.
Mother-child bond | between pregnancy week 36 and 39
  assessement via self-administered questionnaire: Maternal Antenatal Attachment Scale (MAAS) consists of 19 items which are scored 1-5, with higher scores indicating higher levels of bonding.
Sociodemographics | between pregnancy week 9 and 12
  age, education (</=/> school years), partnership, employment status
Left ventricular muscle mass index | Echocardiography between pregnancy week 9 and 12
  Echocardiography will be done by qualified staff.
Left ventricular muscle mass index | cardiac ultrasound measurement between pregnancy week 23 and 26
  Echocardiography will be done by qualified staff.
Left ventricular muscle mass index | Echocardiography between pregnancy week 36 and 39
  Echocardiography will be done by qualified staff.
Echocardiographic global strain, in % | Echocardiography between pregnancy week 9 and 12
  Echocardiography will be done by qualified staff.
Echocardiographic global strain, in % | cardiac ultrasound measurement between pregnancy week 23 and 26
  The cardiac ultrasound examination will be conduced by qualified staff.
Echocardiographic global strain, in % | Echocardiography between pregnancy week 36 and 39
  Echocardiography will be done by qualified staff.

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Ulbricht, Prof., Principal Investigator — University Medicine Greifswald, Dep.Social Medicine and Prevention
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04527731/Prot_000.pdf